CLINICAL TRIAL: NCT03831035
Title: Fast Exome for Diagnosis of Congenital Conditions in Infants Under 12 Months of Age Hospitalized in Intensive Care Unit
Acronym: REUNIR
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0387
Record Dates: First submitted 2019-01-18; First posted 2019-02-05 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Infant, Newborn, Diseases; Congenital Malformations; Intensive Care Unit; Neurologic Symptoms
Keywords: Fast trio exome; Multiple congenital malformation; Intensive care unit; Neurological distress
MeSH Terms: conditions — Infant, Newborn, Diseases; Congenital Abnormalities; Neurologic Manifestations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — It is a trio exome sequencing which includes 3 steps : the analytical step (blood sample DNA extraction and high-throughput sequencing), the bioinformatic step, and the interpretation step.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 15 patients and both parents.: The patients are aged 12 months or under hospitalized in the ICU suffering from multiple congenital malformations and/or neurologic symptoms.
  Interventions: Other: Genetic analyse by whole exome sequencing

INTERVENTIONS:
Other: Genetic analyse by whole exome sequencing — Exome sequencing requires analytic, bio informatic and interpretation steps.

SUMMARY:
An early diagnosis of congenital malformations and suspected genetic conditions in critically ill infants is essential to perform specific adapted care, prevention, and give proper genetic counseling. However, etiologies are various and each of them is individually very rare. Thanks to next-generation sequencing technologies, diagnosis time frames have drastically decreased and the investigators have observed an increase in diagnosis yields.

This study aims to evaluate the feasibility of fast trio exome sequencing (less than 16 days between informed consent signature and the consultation for results to the parents) in infants under the age of 12 months hospitalized in Intensive Care Unit (ICU).

DETAILED DESCRIPTION:
This prospective study is the first French study aiming to evaluate the feasibility of fast trio exome sequencing (less than 16 days between informed consent signature and consultation for results presentation to the parents) in 15 infants under the age of 12 months hospitalized in the Intensive Care Unit. Included patients will have a year of follow-up examination.

The main evaluation criterion is the yield of exome results given to the family before 16 days. The secondary evaluation criteria are 1/ duration of each step until the results 2/ diagnosis yield : identification of the etiology 3/ adjustment of medical care allowed by the exome diagnosis 4/quantity of blood necessary to achieve diagnosis 5/ duration of hospital stay and number of medical consultations in the year following inclusion.

Exome sequencing will be performed on top of classical analysis ordinarily prescribed. Medical care will not be modified until exome results reception. After signature of informed consent, blood samples of the infant and both parents will be used for trio exome sequencing, which includes 3 steps : the analytical step (blood sample DNA extraction and high-throughput sequencing), the bioinformatic step, and the interpretation step.

The study includes four medical consultations:

1/consultation with a geneticist for inclusion, 2/consultation with a geneticist to give the exome results, 3/ consultation at 3 months after the results for the sanger-confirmation of the exome result, 4/ consultation at one year after the inclusion for medical follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Infant aged under 12 months , hospitalized in the ICU.
* Infant with multiple congenital malformations or neurological symptoms for which a genetic origin is suspected but undiagnosed genetically.
* Infant for whom both biological parents have given consent for the study, genetic analysis for themselves anf their child.
* Infant and parents registered in the French National health service

Exclusion Criteria:

* Absence of one or both parental sample.
* Precise genetic diagnosis made pre- or post-natally with chromosomal (I.e : Down syndrome), Sanger (i.e : infantile spinal amyotrophia) methylation (i.e : Prader-Willi syndrome) or triplet amplification (I.e : neonatal Steinert myotonia) studies.
* Strong clinical evidence for a with chromosomal (I.e : Down syndrome), Sanger (i.e : infantile spinal amyotrophia) methylation (i.e : Prader-Willi syndrome) or triplet amplification (I.e : neonatal Steinert myotonia) studies.
* Impossibility for one or both parents to give his or her consent

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study includes 15 patients and both parents. The patients are aged 12 months or under hospitalized in the ICU suffering from multiple congenital malformations and/or neurologic symptoms
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2022-06-08 (Actual)

PRIMARY OUTCOMES:
Yield of exome results given to the family before 16 days | 16 days maximum after inclusion
  number of days between the collect sample and results

SECONDARY OUTCOMES:
Duration of each step until the results (the analytical step, the bioinformatic step, the interpretation step). | 16 days maximum after inclusion
  number of days between the collect sample and results
Diagnosis yield : identification of the etiology | 3 months
  number of days between the collect sample and diagnostic confirmation
Adjustment of medical care allowed by the exome diagnosis | 16 days maximum after inclusion
  Any additions or deletions of a diagnostic exam, medical care specific to the diagnosed pathology or screening of a known complication
Quantity of blood necessary to achieve diagnosis | 16 days maximum after inclusion
  blood volume necessary to achieve diagnosis
Quantity of blood necessary to achieve diagnosis | 16 days maximum after inclusion
  number of samples necessary to achieve diagnosis
duration of hospital stay in the year following inclusion | a year after inclusion
  number of days of hospital stay in the year
number of medical consultations in the year following inclusion | a year after inclusion
  number of medical consultations in the year

CONTACTS AND LOCATIONS:
Overall Officials: Marjolaine WILLEMS, Principal Investigator — Medical genetics Arnaud de Villeneuve
Locations (1):
- Medical genetics Arnaud de Villeneuve, Montpellier, Hérault, France

REFERENCES:
- [Background] Acikalin A, Bagir EK, Torun G, Ates BT, Erdogan S, Uguz A, Ergin M, Buyukkurt S, Ozgunen FT, Tunali N, Gumurdulu D. Perinatal autopsy evaluation of 2150 autopsies in the Cukurova region of Turkey. Turk Patoloji Derg. 2014;30(3):189-94. doi: 10.5146/tjpath.2014.01266. PMID 24994614
- [Background] Baird PA, Anderson TW, Newcombe HB, Lowry RB. Genetic disorders in children and young adults: a population study. Am J Hum Genet. 1988 May;42(5):677-93. PMID 3358420
- [Background] Bonnet D. [Genetics of congenital heart diseases]. Presse Med. 2017 Jun;46(6 Pt 1):612-619. doi: 10.1016/j.lpm.2017.05.014. Epub 2017 Jun 2. French. PMID 28583745
- [Background] Dhiman V. Molecular Genetics of Epilepsy: A Clinician's Perspective. Ann Indian Acad Neurol. 2017 Apr-Jun;20(2):96-102. doi: 10.4103/aian.AIAN_447_16. PMID 28615892
- [Background] Grandemange S, Sanchez E, Louis-Plence P, Tran Mau-Them F, Bessis D, Coubes C, Frouin E, Seyger M, Girard M, Puechberty J, Costes V, Rodiere M, Carbasse A, Jeziorski E, Portales P, Sarrabay G, Mondain M, Jorgensen C, Apparailly F, Hoppenreijs E, Touitou I, Genevieve D. A new autoinflammatory and autoimmune syndrome associated with NLRP1 mutations: NAIAD (NLRP1-associated autoinflammation with arthritis and dyskeratosis). Ann Rheum Dis. 2017 Jul;76(7):1191-1198. doi: 10.1136/annrheumdis-2016-210021. Epub 2016 Dec 13. PMID 27965258
- [Background] Hack M, Taylor HG, Drotar D, Schluchter M, Cartar L, Andreias L, Wilson-Costello D, Klein N. Chronic conditions, functional limitations, and special health care needs of school-aged children born with extremely low-birth-weight in the 1990s. JAMA. 2005 Jul 20;294(3):318-25. doi: 10.1001/jama.294.3.318. PMID 16030276
- [Background] McCandless SE, Brunger JW, Cassidy SB. The burden of genetic disease on inpatient care in a children's hospital. Am J Hum Genet. 2004 Jan;74(1):121-7. doi: 10.1086/381053. Epub 2003 Dec 12. PMID 14681831
- [Background] Musante L, Ropers HH. Genetics of recessive cognitive disorders. Trends Genet. 2014 Jan;30(1):32-9. doi: 10.1016/j.tig.2013.09.008. Epub 2013 Oct 28. PMID 24176302
- [Background] Pabinger S, Dander A, Fischer M, Snajder R, Sperk M, Efremova M, Krabichler B, Speicher MR, Zschocke J, Trajanoski Z. A survey of tools for variant analysis of next-generation genome sequencing data. Brief Bioinform. 2014 Mar;15(2):256-78. doi: 10.1093/bib/bbs086. Epub 2013 Jan 21. PMID 23341494
- [Background] Packer JS, Maxwell EK, O'Dushlaine C, Lopez AE, Dewey FE, Chernomorsky R, Baras A, Overton JD, Habegger L, Reid JG. CLAMMS: a scalable algorithm for calling common and rare copy number variants from exome sequencing data. Bioinformatics. 2016 Jan 1;32(1):133-5. doi: 10.1093/bioinformatics/btv547. Epub 2015 Sep 17. PMID 26382196
- [Background] Richards S, Aziz N, Bale S, Bick D, Das S, Gastier-Foster J, Grody WW, Hegde M, Lyon E, Spector E, Voelkerding K, Rehm HL; ACMG Laboratory Quality Assurance Committee. Standards and guidelines for the interpretation of sequence variants: a joint consensus recommendation of the American College of Medical Genetics and Genomics and the Association for Molecular Pathology. Genet Med. 2015 May;17(5):405-24. doi: 10.1038/gim.2015.30. Epub 2015 Mar 5. PMID 25741868
- [Background] Van der Auwera GA, Carneiro MO, Hartl C, Poplin R, Del Angel G, Levy-Moonshine A, Jordan T, Shakir K, Roazen D, Thibault J, Banks E, Garimella KV, Altshuler D, Gabriel S, DePristo MA. From FastQ data to high confidence variant calls: the Genome Analysis Toolkit best practices pipeline. Curr Protoc Bioinformatics. 2013;43(1110):11.10.1-11.10.33. doi: 10.1002/0471250953.bi1110s43. PMID 25431634
- [Background] Vissers LE, Gilissen C, Veltman JA. Genetic studies in intellectual disability and related disorders. Nat Rev Genet. 2016 Jan;17(1):9-18. doi: 10.1038/nrg3999. Epub 2015 Oct 27. PMID 26503795
- [Background] Zlotogora J, Shalev SA. The consequences of consanguinity on the rates of malformations and major medical conditions at birth and in early childhood in inbred populations. Am J Med Genet A. 2010 Aug;152A(8):2023-8. doi: 10.1002/ajmg.a.33537. PMID 20635393
- [Result] Cunniff C, Carmack JL, Kirby RS, Fiser DH. Contribution of heritable disorders to mortality in the pediatric intensive care unit. Pediatrics. 1995 May;95(5):678-81. PMID 7724302
- [Result] FitzPatrick DR, Skeoch CH, Tolmie JL. Genetic aspects of admissions to a paediatric intensive care unit. Arch Dis Child. 1991 May;66(5):639-41. doi: 10.1136/adc.66.5.639. PMID 2039259
- [Result] Gilissen C, Hoischen A, Brunner HG, Veltman JA. Unlocking Mendelian disease using exome sequencing. Genome Biol. 2011 Sep 14;12(9):228. doi: 10.1186/gb-2011-12-9-228. PMID 21920049
- [Result] Hildreth A, Wigby K, Chowdhury S, Nahas S, Barea J, Ordonez P, Batalov S, Dimmock D, Kingsmore S; RCIGM Investigators. Rapid whole-genome sequencing identifies a novel homozygous NPC1 variant associated with Niemann-Pick type C1 disease in a 7-week-old male with cholestasis. Cold Spring Harb Mol Case Stud. 2017 Sep 1;3(5):a001966. doi: 10.1101/mcs.a001966. Print 2017 Sep. PMID 28550066
- [Result] Kingsmore SF, Petrikin J, Willig LK, Guest E. Emergency medical genomes: a breakthrough application of precision medicine. Genome Med. 2015 Jul 30;7(1):82. doi: 10.1186/s13073-015-0201-z. eCollection 2015. PMID 26229553
- [Result] Lalani SR. Current Genetic Testing Tools in Neonatal Medicine. Pediatr Neonatol. 2017 Apr;58(2):111-121. doi: 10.1016/j.pedneo.2016.07.002. Epub 2016 Sep 28. PMID 28277305
- [Result] Lee H, Deignan JL, Dorrani N, Strom SP, Kantarci S, Quintero-Rivera F, Das K, Toy T, Harry B, Yourshaw M, Fox M, Fogel BL, Martinez-Agosto JA, Wong DA, Chang VY, Shieh PB, Palmer CG, Dipple KM, Grody WW, Vilain E, Nelson SF. Clinical exome sequencing for genetic identification of rare Mendelian disorders. JAMA. 2014 Nov 12;312(18):1880-7. doi: 10.1001/jama.2014.14604. PMID 25326637
- [Result] Petrikin JE, Willig LK, Smith LD, Kingsmore SF. Rapid whole genome sequencing and precision neonatology. Semin Perinatol. 2015 Dec;39(8):623-31. doi: 10.1053/j.semperi.2015.09.009. Epub 2015 Oct 29. PMID 26521050
- [Result] Reardon S. Fast genetic sequencing saves newborn lives. Nature. 2014 Oct 2;514(7520):13-4. doi: 10.1038/514013a. No abstract available. PMID 25279893
- [Result] Saunders CJ, Miller NA, Soden SE, Dinwiddie DL, Noll A, Alnadi NA, Andraws N, Patterson ML, Krivohlavek LA, Fellis J, Humphray S, Saffrey P, Kingsbury Z, Weir JC, Betley J, Grocock RJ, Margulies EH, Farrow EG, Artman M, Safina NP, Petrikin JE, Hall KP, Kingsmore SF. Rapid whole-genome sequencing for genetic disease diagnosis in neonatal intensive care units. Sci Transl Med. 2012 Oct 3;4(154):154ra135. doi: 10.1126/scitranslmed.3004041. PMID 23035047
- [Result] Smith LD, Willig LK, Kingsmore SF. Whole-Exome Sequencing and Whole-Genome Sequencing in Critically Ill Neonates Suspected to Have Single-Gene Disorders. Cold Spring Harb Perspect Med. 2015 Dec 18;6(2):a023168. doi: 10.1101/cshperspect.a023168. PMID 26684335
- [Result] Soden SE, Saunders CJ, Willig LK, Farrow EG, Smith LD, Petrikin JE, LePichon JB, Miller NA, Thiffault I, Dinwiddie DL, Twist G, Noll A, Heese BA, Zellmer L, Atherton AM, Abdelmoity AT, Safina N, Nyp SS, Zuccarelli B, Larson IA, Modrcin A, Herd S, Creed M, Ye Z, Yuan X, Brodsky RA, Kingsmore SF. Effectiveness of exome and genome sequencing guided by acuity of illness for diagnosis of neurodevelopmental disorders. Sci Transl Med. 2014 Dec 3;6(265):265ra168. doi: 10.1126/scitranslmed.3010076. PMID 25473036
- [Result] Thevenon J, Duffourd Y, Masurel-Paulet A, Lefebvre M, Feillet F, El Chehadeh-Djebbar S, St-Onge J, Steinmetz A, Huet F, Chouchane M, Darmency-Stamboul V, Callier P, Thauvin-Robinet C, Faivre L, Riviere JB. Diagnostic odyssey in severe neurodevelopmental disorders: toward clinical whole-exome sequencing as a first-line diagnostic test. Clin Genet. 2016 Jun;89(6):700-7. doi: 10.1111/cge.12732. Epub 2016 Apr 26. PMID 26757139
- [Result] Willig LK, Petrikin JE, Smith LD, Saunders CJ, Thiffault I, Miller NA, Soden SE, Cakici JA, Herd SM, Twist G, Noll A, Creed M, Alba PM, Carpenter SL, Clements MA, Fischer RT, Hays JA, Kilbride H, McDonough RJ, Rosterman JL, Tsai SL, Zellmer L, Farrow EG, Kingsmore SF. Whole-genome sequencing for identification of Mendelian disorders in critically ill infants: a retrospective analysis of diagnostic and clinical findings. Lancet Respir Med. 2015 May;3(5):377-87. doi: 10.1016/S2213-2600(15)00139-3. Epub 2015 Apr 27. PMID 25937001
- [Result] Yang Y, Muzny DM, Reid JG, Bainbridge MN, Willis A, Ward PA, Braxton A, Beuten J, Xia F, Niu Z, Hardison M, Person R, Bekheirnia MR, Leduc MS, Kirby A, Pham P, Scull J, Wang M, Ding Y, Plon SE, Lupski JR, Beaudet AL, Gibbs RA, Eng CM. Clinical whole-exome sequencing for the diagnosis of mendelian disorders. N Engl J Med. 2013 Oct 17;369(16):1502-11. doi: 10.1056/NEJMoa1306555. Epub 2013 Oct 2. PMID 24088041